CLINICAL TRIAL: NCT00518180
Title: A Phase 3, Single-Center, Open-label, Controlled, Randomized Study to Evaluate the Safety and Immunogenicity of Novartis Men ACWY Vaccine Administered Either Alone or Concomitantly With a Combined Tetanus, Reduced Diphtheria Toxoid, Acellular Pertussis Vaccine and Quadrivalent Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine in Healthy Adolescents
Brief Title: A Study to Evaluate Safety and Immune Response of Novartis Meningococcal ACWY Conjugate Vaccine In Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P18
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Results first posted 2010-10-04 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Meningococcal Meningitis; Human Papillomavirus Infection; Pertussis; Tetanus
Keywords: Meningococcal; meningitis; vaccine; adolescents
MeSH Terms: conditions — Meningitis, Meningococcal; Papillomavirus Infections; Whooping Cough; Tetanus; Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MenACWY + Tdap + HPV (Experimental): Subjects received MenACWY concomitantly with Tdap and HPV at study month 0 followed by two injections of HPV at month 2 and 6
  Interventions: Biological: Novartis Meningococcal ACWY Conjugate Vaccine
- MenACWY →Tdap → HPV (Experimental): Subjects received MenACWY at study month 0 followed by one injection of Tdap at month 1, followed by three injections of HPV at months 2, 4, and 8
  Interventions: Biological: Novartis Meningococcal ACWY Conjugate Vaccine
- Tdap →MenACWY → HPV (Experimental): Subjects received Tdap at month 0 followed by one injection of MenACWY at month 1, followed by three injections of HPV at months 2, 4, and 8
  Interventions: Biological: Tdap Vaccine

INTERVENTIONS:
Biological: Novartis Meningococcal ACWY Conjugate Vaccine — One dose of vaccine administered intramuscularly
  Arms: MenACWY + Tdap + HPV
Biological: Tdap Vaccine — One dose of vaccine administered intramuscularly
  Arms: Tdap →MenACWY → HPV
Biological: Novartis Meningococcal ACWY Conjugate Vaccine — One dose of vaccine administered intramuscularly
  Arms: MenACWY →Tdap → HPV

SUMMARY:
This study will evaluate the safety and immune response of the Novartis Meningococcal ACWY conjugate vaccine when administered with Tdap and HPV vaccinations to healthy adolescents

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents 11-18 years of age
* virgins (both male and female) with no intention of becoming sexually active during the study period
* who have been properly vaccinated against diphtheria, tetanus, pertussis

Exclusion Criteria:

* who had a previous confirmed or suspected disease caused by N. meningitidis;
* who have previously been immunized with a meningococcal vaccine
* who have received prior human papillomavirus (HPV) vaccine;
* who have any serious acute, chronic or progressive disease
* who have epilepsy, any progressive neurological disease or history of Guillain-Barre syndrome;
* who have a known or suspected impairment/alteration of immune function, either congenital or acquired
* who are known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
* who have Down's syndrome or other known cytogenic disorders;

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1620 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (1):
- San Jose, Costa Rica, San José, Costa Rica

REFERENCES:
- [Result] Arguedas A, Soley C, Loaiza C, Rincon G, Guevara S, Perez A, Porras W, Alvarado O, Aguilar L, Abdelnour A, Grunwald U, Bedell L, Anemona A, Dull PM. Safety and immunogenicity of one dose of MenACWY-CRM, an investigational quadrivalent meningococcal glycoconjugate vaccine, when administered to adolescents concomitantly or sequentially with Tdap and HPV vaccines. Vaccine. 2010 Apr 19;28(18):3171-9. doi: 10.1016/j.vaccine.2010.02.045. Epub 2010 Feb 26. PMID 20189491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a single center in Costa Rica.
Pre-assignment Details: All enrolled subjects were randomized at a 1:1:1 ratio to receive the MenACWY vaccine when given alone and concomitantly with the Tdap vaccine and the HPV vaccine at different schedules.
Groups:
- MenACWY+Tdap+HPV: The MenACWY vaccine was administered concomitantly with the Tdap vaccine and the HPV vaccine at study month 0 followed by two injections of the HPV vaccine at months 2 and 6.
- MenACWY→Tdap→HPV: The MenACWY vaccine was administered at study month 0 followed by one injection of the Tdap vaccine at month 1, followed by three injections of the HPV vaccine at months 2, 4, and 8.
- Tdap →MenACWY → HPV: Tdap vaccine was administered at month 0 followed by one injection of MenACWY at month 1, followed by three injections of the HPV vaccine at months 2, 4, and 8.
Period: Overall Study
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap →MenACWY → HPV
Started | 540 | 541 | 539
Completed | 475 | 472 | 457
Not Completed | 65 | 69 | 82
Not completed — Withdrawal by Subject | 29 | 30 | 42
Not completed — Lost to Follow-up | 30 | 28 | 34
Not completed — Administrative reason | 0 | 2 | 2
Not completed — Protocol Violation | 5 | 7 | 4
Not completed — Unable to classify | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap →MenACWY → HPV | Total
Number analyzed (Participants) | 540 | 541 | 539 | 1620
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (2.1) | 13.9 (2.2) | 13.8 (2.2) | 13.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 309 | 307 | 924
  Male | 232 | 232 | 232 | 696
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 539 | 541 | 539 | 1619
  Black | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Human Serum Bactericidal Assay (hSBA) Seroresponse
Description: Immune responses to MenACWY, as measured by the percentage of hSBA seroresponders, when given: (a) alone; (b) concomitantly with a Tetanus diphtheria acellular pertussis (Tdap) vaccine and a Human Papillomavirus Recombinant (HPV) vaccine; and (c) when given one month after a Tdap vaccine.
  Seroresponse to MenACWY: For a subject with baseline hSBA titer <1:4, seroresponse is defined as a postvaccination hSBA titer ≥ 1:8; for a subject with baseline hSBA titer ≥ 1:4, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 1 month post MenACWY vaccination
Population: The analysis was performed on the per-protocol (PP) population. A total of 182 subjects were excluded from the PP population due to protocol deviations. The most common protocol deviations were blood draw performed outside the protocol-specified window.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap →MenACWY → HPV
Number analyzed (Participants) | 494 | 487 | 458
Percentage of participants
  Serogroup A (N=494, 486, 458) | 80 [76 to 84] | 82 [78 to 85] | 87 [83 to 90]
  Serogroup C (N=476, 472, 457) | 83 [79 to 86] | 84 [81 to 88] | 84 [80 to 87]
  Serogroup W (N=487, 474, 458) | 77 [73 to 80] | 81 [77 to 84] | 65 [61 to 70]
  Serogroup Y (N=493, 487, 460) | 83 [79 to 86] | 82 [79 to 86] | 78 [74 to 82]
Statistical Analysis 1: Comparison: MenACWY+Tdap+HPV vs MenACWY→Tdap→HPV; Immune response to Men A when MenACWY is administered concomitantly with Tdap and HPV, compared with the immune response to MenACWY when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — The immunogenicity of MenACWY given concomitantly with HPV and Tdap was considered non inferior to the immunogenicity of MenACWY administered alone, if, for each serogroup, the lower limit of the two-sided 95% confidence interval (CI) for the difference in percentage of subjects with seroresponse at one month after MenACWY vaccination (PGroup I minus PGroup II) was greater than -10%; Vaccine Group differences (%) = -2, 95% CI 2-sided [-6 to 3]
Statistical Analysis 2: Comparison: MenACWY+Tdap+HPV vs MenACWY→Tdap→HPV; Immune response to Men C when MenACWY is administered concomitantly with Tdap and HPV, compared with the immune response to MenACWY when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Vaccine Group differences (%) = -1, 95% CI 2-sided [-6 to 3]
Statistical Analysis 3: Comparison: MenACWY+Tdap+HPV vs MenACWY→Tdap→HPV; Immune response to Men W when MenACWY is administered concomitantly with Tdap and HPV, compared with the immune response to MenACWY when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Vaccine Group differences (%) = -4, 95% CI 2-sided [-9 to 1]
Statistical Analysis 4: Comparison: MenACWY+Tdap+HPV vs MenACWY→Tdap→HPV; Immune response to Men Y when MenACWY is administered concomitantly with Tdap and HPV, compared with the immune response to MenACWY when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Vaccine Group differences (%) = 0, 95% CI 2-sided [-4 to 5]
Statistical Analysis 5: Comparison: MenACWY→Tdap→HPV vs Tdap →MenACWY → HPV; Immune response to Men A when MenACWY is administered 1 month after Tdap, compared with the immune response to MenACWY when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — The immunogenicity of MenACWY given after Tdap was considered non inferior to the immunogenicity of MenACWY administered alone, if, for each serogroup, the lower limit of the two-sided 95% confidence interval (CI) for the difference in percentage of subjects with seroresponse at one month after MenACWY vaccination (PGroup III minus PGroup II) was greater than -10%; Vaccine Group differences (%) = 5, 95% CI 2-sided [1 to 10]
Statistical Analysis 6: Comparison: MenACWY→Tdap→HPV vs Tdap →MenACWY → HPV; Immune response to Men C when MenACWY is administered 1 month after Tdap, compared with the immune response to MenACWY when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 5]; Vaccine Group differences (%) = -1, 95% CI 2-sided [-6 to 4]
Statistical Analysis 7: Comparison: MenACWY→Tdap→HPV vs Tdap →MenACWY → HPV; Immune response to Men W when MenACWY is administered 1 month after Tdap, compared with the immune response to MenACWY when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 5]; Vaccine Group differences (%) = -16, 95% CI 2-sided [-21 to -10]
Statistical Analysis 8: Comparison: MenACWY→Tdap→HPV vs Tdap →MenACWY → HPV; Immune response to Men Y when MenACWY is administered 1 month after Tdap, compared with the immune response to MenACWY when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 5]; Vaccine Group differences (%) = -4, 95% CI 2-sided [-9 to 1]

2. Primary Outcome: Percentage of Subjects With Antidiphtheria and Antitetanus Toxin ≥1.0 IU/mL
Description: To compare the immune response to Tdap given concomitantly with MenACWY and HPV vaccine with the immune response to Tdap when administered alone
Time Frame: 1 month post Tdap vaccination
Population: The analysis was performed on the per-protocol (PP) population. A total of 183 subjects were excluded from the PP population due to protocol deviations. The most common protocol deviations were blood draw performed outside the protocol-specified window.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap →MenACWY → HPV
Number analyzed (Participants) | 492 | 458 | 487
Percentage of subjects
  Diphtheria | 100 [99 to 100] | 100 [99 to 100] | 98 [96 to 99]
  Tetanus | 100 [99 to 100] | 100 [99 to 100] | 100 [99 to 100]
Statistical Analysis 1: Comparison: MenACWY+Tdap+HPV vs Tdap →MenACWY → HPV; Non inferiority of the immune response to diphteria antigen, when Tdap is administered concomitantly with MenACWY and HPV, compared with the immune response to Tdap when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — Non inferiority of the immune response to Tdap when administered concomitantly with MenACWY and HPV, compared with the immune response to Tdap when administered alone, was demonstrated for the diphteria and tetanus antigens if the lower limits of the two-sided 95% CIs around the difference in the percentages of subjects with ELISA anti-D toxin ≥ 1.0 IU/mL [Group I minus Group III] were greater than -10%; Vaccine Group differences (%) = 2, 95% CI 2-sided [1 to 4]
Statistical Analysis 2: Comparison: MenACWY+Tdap+HPV vs Tdap →MenACWY → HPV; Non inferiority of the immune response to tetanus antigen, when Tdap is administered concomitantly with MenACWY and HPV, compared with the immune response to Tdap when administered alone. Method: ANCOVA. Parameter estimate: Vaccine Group Differences; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group differences (%) = 0, 95% CI 2-sided [-1 to 1]

3. Secondary Outcome: Effect of Concomitant and Sequential Vaccination on hSBA Geometric Mean Titers (GMTs) for A, C, W, and Y Serogroups
Description: The immune responses to the MenACWY conjugate vaccine, as measured by the hSBA Geometric Mean Titers (GMTs) when given: (a) alone, (b) concomitantly with the Tdap vaccine and the HPV vaccine, and (c) when given one month after the Tdap vaccine.
Time Frame: 1 month post MenACWY vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Tdap → MenACWY→HPV: Tdap was administered at study month 0 followed by one injection of the MenACWY vaccine at month 1, followed by three injections of the HPV vaccine at months 2, 4, and 8.
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap → MenACWY→HPV
Number analyzed (Participants) | 494 | 487 | 460
Titers
  Serogroup A (N=494, 486, 458) | 62 [52 to 74] | 67 [56 to 80] | 95 [79 to 113]
  Serogroup C (N=476, 472, 457) | 66 [56 to 77] | 70 [60 to 83] | 68 [58 to 79]
  Serogroup W (N=487, 474, 458) | 146 [129 to 165] | 159 [140 to 181] | 104 [91 to 119]
  Serogroup Y (N=493, 487, 460) | 72 [62 to 84] | 81 [70 to 95] | 57 [49 to 67]

4. Secondary Outcome: Percentage of Subjects With Anti-HPV Seroconversion
Description: To compare the immune response of HPV vaccine given concomitantly with MenACWY and Tdap to the response when HPV vaccine is given alone. (Immune response against HPV virus-like particles (VLPs) for types 6, 11, 16, and 18 was measured at one month after the third HPV vaccination.) Anti-HPV Seroconversion (SC): SC was defined as negative (baseline HPV titer < type-specific cut-off) for anti-HPV and anti-HPV ≥ an HPV type-specific cut-off at one month after the third HPV injection.
Time Frame: 1 month post third HPV vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- HPV Alone: Three injections of the HPV vaccine were administered at study months 2, 4, and 8. This arm is a recombination of the two arms listed in the Participant Flow.
Arm/Group | MenACWY+Tdap+HPV | HPV Alone
Number analyzed (Participants) | 364 | 744
Percentage of subjects
  HPV 6 (N=361, 737) | 99 [98 to 100] | 100 [99 to 100]
  HPV 11 (N=362, 744) | 100 [99 to 100] | 100 [99 to 100]
  HPV 16 (N=360, 744) | 100 [99 to 100] | 100 [99 to 100]
  HPV 18 (N=364, 743) | 100 [98 to 100] | 99 [99 to 100]

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Anti-HPV by Competitive Luminex Immunoassay
Description: To compare the immune response of HPV vaccine given concomitantly with MenACWY and Tdap to the response when HPV vaccine is given alone. (Immune response against HPV virus-like particles (VLPs) for types 6, 11, 16, and 18 was measured at one month after the third HPV vaccine vaccination.)
Time Frame: 1 month post third HPV vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- HPV Alone: The three injections of the HPV vaccine was administered at study months 2, 4, and 8. This arm is a recombination of the two arms listed in the Participant Flow.
Arm/Group | MenACWY+Tdap+HPV | HPV Alone
Number analyzed (Participants) | 364 | 745
Titers
  HPV 6 (N=361, 737) | 1059 [926 to 1212] | 1461 [1327 to 1608]
  HPV 11 (N=362, 744) | 1264 [1134 to 1408] | 1701 [1575 to 1837]
  HPV 16 (N=360, 744) | 5286 [4705 to 5939] | 6590 [6068 to 7158]
  HPV 18 (N=364, 743) | 908 [798 to 1032] | 1117 [1019 to 1224]

6. Secondary Outcome: Percentage of Subjects With hSBA ≥ 1:8, hSBA Titer ≥ 1:4, for A, C, W, and Y Serogroups
Description: The immune responses to MenACWY, as measured by the percentage of subjects with hSBA titer ≥ 1:8, hSBA titer ≥ 1:4, when given: (a) alone, (b) concomitantly with Tdap and HPV vaccine; and (c) when given one month after Tdap.
Time Frame: 1 month post MenACWY vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap → MenACWY→HPV
Number analyzed (Participants) | 475 | 472 | 457
Percentage of subjects
  Serogroup A hSBA ≥ 1:8 (N=494, 486, 458) | 81 [78 to 85] | 82 [79 to 86] | 89 [85 to 91]
  Serogroup C hSBA ≥ 1:8 (N=476, 472, 457) | 92 [89 to 94] | 90 [87 to 93] | 93 [90 to 95]
  Serogroup W hSBA ≥ 1:8 (N=487, 474, 458) | 98 [96 to 99] | 99 [98 to 100] | 95 [93 to 97]
  Serogroup Y hSBA ≥ 1:8 (N=493, 487, 460) | 93 [90 to 95] | 93 [90 to 95] | 92 [90 to 95]
  Serogroup A hSBA ≥ 1:4 (N=408, 404, 412) | 83 [79 to 86] | 83 [79 to 86] | 90 [87 to 93]
  Serogroup C hSBA ≥ 1:4 (N=456, 447, 430) | 92 [90 to 94] | 92 [89 to 94] | 94 [92 to 96]
  Serogroup W hSBA ≥ 1:4 (N=478, 471, 443) | 98 [97 to 99] | 99 [98 to 100] | 97 [95 to 98]
  Serogroup Y hSBA ≥ 1:4 (N=465, 456, 438) | 94 [92 to 96] | 94 [91 to 96] | 95 [93 to 97]

7. Secondary Outcome: The Effect of Sequential Vaccination on Immunogenicity for Diphtheria and Tetanus
Description: The immune response to the Tdap vaccine, as measured by the percentage of subjects with antidiphtheria and antitetanus toxin ≥1.0 IU/mL.
Time Frame: 1 month post Tdap vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap → MenACWY→HPV
Number analyzed (Participants) | 492 | 458 | 487
Percentages of subjects
  Diphtheria (% ≥1.0 IU/mL) | 100 [99 to 100] | 100 [99 to 100] | 98 [96 to 99]
  Tetanus (% ≥1.0 IU/mL) | 100 [99 to 100] | 100 [99 to 100] | 100 [99 to 100]

8. Secondary Outcome: Geometric Mean Concentrations (GMC) for Diphtheria and Tetanus
Description: To compare the immune response of Tdap, as measured by the antidiphtheria and antitetanus GMCs, when administered one month after the MenACWY vaccine with the immune response of the Tdap vaccine when administered alone.
Time Frame: 1 month post Tdap vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap → MenACWY→HPV
Number analyzed (Participants) | 492 | 458 | 487
IU/mL
  Diphtheria | 37 [34 to 41] | 10 [9.12 to 12] | 10 [9.38 to 11]
  Tetanus | 8.75 [8.23 to 9.3] | 12 [11 to 13] | 10 [9.46 to 11]

9. Secondary Outcome: Geometric Mean Titers (GMT) of Pertussis Antigens
Description: To compare the immune response to Tdap administered one month after MenACWY with the immune response to Tdap administered alone.
Time Frame: 1 month post Tdap vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap → MenACWY→HPV
Number analyzed (Participants) | 492 | 458 | 487
Titers
  Anti-PT (N=479, 451, 477) | 51 [47 to 55] | 79 [72 to 87] | 63 [58 to 69]
  Anti-FHA (N=489, 457, 485) | 342 [310 to 376] | 1106 [989 to 1238] | 511 [464 to 563]
  Anti-PRN (N=492, 458, 487) | 819 [727 to 923] | 1563 [1390 to 1758] | 1197 [1061 to 1350]

10. Secondary Outcome: Percentages of Subjects With at Least a 4-fold Rise for PT, FHA, and PRN
Description: To compare the immune response of Tdap, defined by the percentage of subjects with a 4-fold rise in antibody titer over baseline against PT, FHA, PRN, when administered one month after the MenACWY with the immune response of Tdap when administered alone.
Time Frame: 1 month post Tdap vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap → MenACWY→HPV
Number analyzed (Participants) | 492 | 458 | 487
Percentages of subjects
  Anti-PT (N=479, 451, 477) | 83 [79 to 86] | 89 [86 to 92] | 86 [83 to 89]
  Anti-FHA (N=489, 457, 485) | 67 [63 to 71] | 90 [87 to 93] | 78 [74 to 82]
  Anti-PRN (N=492, 458, 487) | 86 [83 to 89] | 95 [92 to 97] | 89 [85 to 91]

11. Primary Outcome: Geometric Mean Concentrations (GMC) of Antipertussis Toxin (Anti-PT), Antifilamentous Hemagglutinin (Anti-FHA), and Antipertactin (Anti-PRN)
Description: To compare the immune response of Tdap given concomitantly with MenACWY and HPV vaccine with the immune response of Tdap when administered alone
Time Frame: 1 month post Tdap vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap →MenACWY → HPV
Number analyzed (Participants) | 492 | 458 | 487
IU/mL
  Anti-PT (N=479, 451, 477) | 51 [47 to 55] | 79 [72 to 87] | 63 [58 to 69]
  Anti-FHA (N=489, 457, 485) | 342 [310 to 376] | 1106 [989 to 1238] | 511 [464 to 563]
  Anti-PRN (N=492, 458, 487) | 819 [727 to 923] | 1563 [1390 to 1758] | 1197 [1061 to 1350]
Statistical Analysis 1: Comparison: MenACWY+Tdap+HPV vs Tdap →MenACWY → HPV; Non inferiority of the immune response to Tdap is administered concomitantly with MenACWY and HPV, compared with the immune response to Tdap when administered alone, for PT antigen. Method: ANCOVA. Parameter estimate: Vaccine Group Ratio; Test type: Non-Inferiority or Equivalence — Tdap concomitant with MenACWY a was considered non inferior to Tdap alone if, for PT, FHA and pertactin, the lower limit of the two-sided 95% CI for the ratio of the GMCs (GMC Group I / GMC Group III) at 1 month after vaccination was > 0.67; Vaccine Group Ratio = 0.8, 95% CI 2-sided [0.72 to 0.9]
Statistical Analysis 2: Comparison: MenACWY+Tdap+HPV vs Tdap →MenACWY → HPV; Non inferiority of the immune response to Tdap when administered concomitantly with MenACWY and HPV, compared with the immune response to Tdap when administered alone, for PRN antigen. Method: ANCOVA. Parameter estimate: Vaccine Group Ratio; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 11, analysis 1]; Vaccine Group Ratio = 0.68, 95% CI 2-sided [0.58 to 0.81]
Statistical Analysis 3: Comparison: MenACWY+Tdap+HPV vs Tdap →MenACWY → HPV; Non inferiority of the immune response to Tdap when administered concomitantly with MenACWY and HPV, compared with the immune response to Tdap when administered alon, for FHA antigen. Method: ANCOVA. Parameter estimate: Vaccine Group Ratio; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 11, analysis 1]; Vaccine Group Ratio = 0.67, 95% CI 2-sided [0.58 to 0.76]

12. Secondary Outcome: Number of Subjects With at Least One Reactogenicity Sign After MenACWY and Tdap Vaccination.
Description: Number of subjects with specified local and systemic reactions were assessed when MenACWY was given alone, one month after Tdap, and concomitantly with Tdap and HPV vaccine.
Time Frame: Days 1 to 7
Population: The analysis was performed on the safety set.
Measure: Number; unit: Subjects
Groups:
- MenACWY→Tdap → HPV: The MenACWY vaccine was administered at study month 0 followed by one injection of the Tdap vaccine at month 1, followed by three injections of the HPV vaccine at months 2, 4, and 8.
- Tdap → MenACWY →HPV: Tdap vaccine was administered at month 0 followed by one injection of MenACWY at month 1, followed by three injections of the HPV vaccine at months 2, 4, and 8.
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap → HPV | Tdap → MenACWY →HPV
Number analyzed (Participants) | 540 | 541 | 539
Subjects
  Injection site pain MenACWY | 263 | 246 | 239
  Injection site pain Tdap | 367 | 310 | 383
  Injection site erythema MenACWY | 68 | 66 | 64
  Injection site erythema Tdap | 78 | 38 | 70
  Injection site induration MenACWY | 68 | 70 | 63
  Injection site induration Tdap | 90 | 64 | 110
  Chills post-vaccination 1 | 77 | 66 | 70
  Chills post-vaccination 2 | 0 | 42 | 45
  Nausea post-vaccination 1 | 88 | 72 | 82
  Nausea post-vaccination 2 | 0 | 42 | 64
  Malaise post-vaccination 1 | 133 | 110 | 115
  Malaise post-vaccination 2 | 0 | 91 | 88
  Myalgia post-vaccination 1 | 146 | 104 | 142
  Myalgia post-vaccination 2 | 0 | 81 | 82
  Arthralgia post-vaccination 1 | 94 | 62 | 76
  Arthralgia post-vaccination 2 | 0 | 52 | 52
  Headache post-vaccination 1 | 217 | 194 | 200
  Headache post-vaccination 2 | 0 | 125 | 138
  Rash post-vaccination 1 | 21 | 17 | 20
  Rash post-vaccination 2 | 0 | 15 | 13
  Fever ≥ 38°Celsius post-vaccination 1 | 27 | 19 | 17
  Fever ≥ 38°Celsius post-vaccination 2 | 0 | 25 | 30
  Analgesic/Antipyretic Med. Used post-vaccination 1 | 110 | 83 | 96
  Analgesic/Antipyretic Med. Used post-vaccination 2 | 0 | 58 | 49

13. Secondary Outcome: Number of Subjects With at Least One Reactogenicity Sign After Each HPV Vaccination
Description: Number of subjects with specified local and systemic reactions were solicited for 7 days after the HPV vaccination.
Time Frame: Days 1 to 7
Population: The analysis was performed on the safety population.
Measure: Number; unit: Subjects
Groups:
- MenACWY+Tdap+HPV: The MenACWY vaccine was administered concomitantly with the Tdap vaccine and the HPV vaccine at study month 0 followed by two vaccinations of the HPV vaccine at month 2 and 6.
- MenACWY→Tdap→HPV: The MenACWY vaccine was administered at study month 0 followed by one injection of the Tdap vaccine at month 1, followed by three injections of the HPV at months 2, 4, and 8
- Tdap → MenACWY → HPV: Tdap vaccine was administered at month 0 followed by one injection of MenACWY at month 1, followed by three injections of HPV at months 2, 4, and 8
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap → MenACWY → HPV
Number analyzed (Participants) | 540 | 494 | 486
Subjects
  Injection site pain postvaccination 1 | 265 | 180 | 204
  Injection site erythema postvaccination 1 | 74 | 36 | 42
  Injection site induration postvaccination 1 | 54 | 27 | 26
  Injection site pain (N=498, 483, 468) postvac 2 | 208 | 208 | 189
  Injection site erythema postvaccination 2 | 62 | 48 | 57
  Injection site induration postvaccination 2 | 46 | 37 | 50
  Injection site pain postvaccination 3 | 229 | 227 | 208
  Injection site erythema postvaccination 3 | 60 | 56 | 55
  Injection site induration postvaccination 3 | 60 | 47 | 48
  Chills postvaccination 1 | 77 | 27 | 30
  Nausea postvaccination 1 | 88 | 39 | 32
  Malaise postvaccination 1 | 133 | 49 | 55
  Myalgia postvaccination 1 | 146 | 32 | 56
  Arthralgia postvaccination 1 | 94 | 33 | 28
  Headache postvaccination 1 | 217 | 93 | 97
  Rash postvaccination 1 | 21 | 7 | 6
  Fever (≥ 38°C) postvaccination 1 | 27 | 21 | 23
  Stayed home postvaccination 1 | 110 | 26 | 34
  Chills postvaccination 2 | 23 | 22 | 26
  Nausea postvaccination 2 | 38 | 30 | 29
  Malaise postvaccination 2 | 53 | 45 | 34
  Myalgia postvaccination 2 | 42 | 38 | 51
  Arthralgia postvaccination 2 | 30 | 28 | 21
  Headache postvaccination 2 | 88 | 78 | 71
  Rash postvaccination 2 | 4 | 11 | 9
  Fever (≥ 38°C) postvaccination 2 | 17 | 22 | 22
  Chills postvaccination 3 | 22 | 24 | 25
  Nausea postvaccination 3 | 32 | 35 | 34
  Malaise postvaccination 3 | 49 | 50 | 41
  Myalgia postvaccination 3 | 53 | 49 | 37
  Arthralgia postvaccination 3 | 37 | 26 | 30
  Headache postvaccination 3 | 79 | 85 | 79
  Rash postvaccination 3 | 9 | 7 | 10
  Fever (≥ 38°C) postvaccination 3 | 20 | 16 | 25

ADVERSE EVENTS:
Time Frame: During the 30-day period following each vaccination.
Description: Data provided in Other Adverse Events (>5%) were collected during the 7-day period after each vaccination.
Groups:
- MenACWY→Tdap→HPV: The MenACWY vaccine was administered at study month 0 followed by one injection of the Tdpa vaccine at month 1, followed by three injections of the HPV at months 2,4 and 8.
- Tdap → MenACWY → HPV: Tdpa was administered at month 0 followed by one injection of MenACWY at month 1, followed by three injections of HPV at months 2,4 and 8.
Arm/Group | MenACWY+Tdap+HPV | MenACWY→Tdap→HPV | Tdap → MenACWY → HPV
Serious Adverse Events (participants affected / at risk) | 1/540 | 7/541 | 3/539
Other Adverse Events (participants affected / at risk) | 495/540 | 489/541 | 482/539
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY+Tdap+HPV (N=540) | MenACWY→Tdap→HPV (N=541) | Tdap → MenACWY → HPV (N=539)
CUSHING'S SYNDROME (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
BEZOAR (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGIC OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
TESTICULAR TORSION (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
BEHCET'S SYNDROME (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY+Tdap+HPV (N=540) | MenACWY→Tdap→HPV (N=541) | Tdap → MenACWY → HPV (N=539)
NAUSEA (Gastrointestinal disorders) | 124 (191) | 133 (255) | 142 (289)
CHILLS (General disorders) | 100 (131) | 117 (201) | 130 (238)
INJECTION SITE ERYTHEMA HPV (General disorders) | 134 (212) | 105 (147) | 101 (166)
INJECTION SITE INDURATION HPV (General disorders) | 119 (179) | 81 (116) | 85 (134)
INJECTION SITE PAIN HPV (General disorders) | 387 (778) | 320 (666) | 313 (648)
MALAISE (General disorders) | 171 (284) | 209 (402) | 194 (428)
PYREXIA (General disorders) | 62 (77) | 88 (129) | 84 (123)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 119 (188) | 132 (225) | 131 (248)
MYALGIA (Musculoskeletal and connective tissue disorders) | 178 (276) | 187 (339) | 200 (440)
HEADACHE (Nervous system disorders) | 260 (519) | 284 (749) | 278 (802)
RASH (Skin and subcutaneous tissue disorders) | 31 (36) | 47 (64) | 42 (66)
INJECTION SITE ERYTHEMA MENVEO (General disorders) | 69 (80) | 66 (68) | 65 (71)
INJECTION SITE ERYTHEMA Tdap (General disorders) | 78 (93) | 38 (40) | 72 (82)
INJECTION SITE INDURATION MENVEO (General disorders) | 68 (76) | 70 (72) | 65 (68)
INJECTION SITE INDURATION Tdap (General disorders) | 90 (101) | 64 (67) | 110 (125)
INJECTION SITE PAIN MENVEO (General disorders) | 264 (307) | 246 (289) | 239 (266)
INJECTION SITE PAIN Tdap (General disorders) | 368 (407) | 310 (343) | 383 (427)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No